CLINICAL TRIAL: NCT01705366
Title: Clinical Outcomes of Joint Arthroplasty
Brief Title: Clinical Outcomes of Knee Replacement
Status: Terminated | Type: Observational
Why Stopped: Changes in funding.
Sponsor: Northwest Surgical Specialists, Vancouver (Other)
Collaborators: Stryker MAKO Surgical Corp (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAKO-01; Borus 2015-005 (Other: Stryker)
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Knee Arthroplasty
Keywords: Osteoarthritis; Joint Disease; Arthritis; Musculoskeletal Disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Arthritis; Musculoskeletal Diseases | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Arthroplasty: Patients undergoing total knee arthroplasty. This may be Non-MAKO® Robot Assisted Total Knee Arthroplasty or MAKO® Robot Assisted Medial Knee Arthroplasty or MAKO® Robot Assisted Medial and PF Knee Arthroplasty
  The Non-MAKO® Robot Assisted Total Knee Arthroplasty uses the Depuy Knee Replacement System or the Stryker® Knee Replacement System. The MAKO® Robot Assisted Arthroplasty uses the RESTORIS Multicompartmental Knee System .
  Interventions: Procedure: Non-MAKO® Robot Assisted Total Knee Arthroplasty; Procedure: MAKO® Robot Assisted Medial Knee Arthroplasty; Procedure: MAKO® Robot Assisted Medial and PF Knee Arthroplasty; Device: RESTORIS Multicompartmental Knee System; Device: Depuy Knee Replacement System; Device: Stryker® Knee Replacement System

INTERVENTIONS:
Procedure: Non-MAKO® Robot Assisted Total Knee Arthroplasty — Patients undergoing a non-MAKO® robot assisted surgery to replace one or more compartments of the knee.
  Other Names: TKA; Total Knee Replacement; Revision Knee Arthroplasty
Procedure: MAKO® Robot Assisted Medial Knee Arthroplasty — Patients undergoing a MAKO® robot assisted surgery to replace the medial compartment of the knee.
  Other Names: Unicompartmental Knee Arthroplasty (UKA)
Procedure: MAKO® Robot Assisted Medial and PF Knee Arthroplasty — Patients undergoing a MAKO® robot assisted surgery to replace the medial and patellofemoral (PF) compartments of the knee
  Other Names: Bi-compartmental Knee Arthroplasty
Device: RESTORIS Multicompartmental Knee System — The RESTORIS Multicompartmental Knee (MCK) System components are intended for single or multicompartmental knee replacement used in conjunction with the MAKO® Robotic Arm Interactive Orthopedic System (RIO®). The components can be used for medial compartment, lateral compartment, patellofemoral compartment, or bicompartmental (medial and patellofemoral compartments) knee replacement. The device is intended to be used with bone cement.
  Other Names: RESTORIS® MCK MultiCompartmental Knee System; FDA 501K number K090763
Device: Depuy Knee Replacement System — The Depuy Knee Replacement System components are intended for use in total knee replacement. These components are intended for implantation with bone cement.
Device: Stryker® Knee Replacement System — The Stryker® Knee Replacement System components are intended for use in total knee replacement. These components are intended for implantation with bone cement.

SUMMARY:
The objective of this study is to document the demographic and clinical characteristics and the long-term clinical outcomes of patients who require a robot assisted knee arthroplasty.

The hypothesis is that MAKO® robot assisted surgery replacing one or two compartments of the knee joint has 10 year implant survival and clinical outcomes that are equivalent to other knee replacement systems.

ELIGIBILITY:
Inclusion Criteria:

* requires either primary or revision knee replacement surgery because of pain and joint stiffness that interferes with performance of normal daily activities
* has failed non-operative management of their joint disease

Exclusion Criteria:

* cognitively unable to complete study health-related quality of life forms
* pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and non-pregnant females undergoing knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2012-10; Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Survivorship of Components | 10 years
  Survivorship of components is defined as knee implant device(s) remaining in patient.

SECONDARY OUTCOMES:
American Knee Society Knee Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year, 2 years, 5 years, and 10 years after surgery
  The American Knee Society Score is an assessment and questionnaire that provides a rating of the pain, function, range of motion, and knee joint stability. It is subdivided into a knee score that rates only the knee joint itself and a functional score that rates the patient's ability to walk and climb stairs.

OTHER OUTCOMES:
Reduced WOMAC | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year, 2 years, 5 years, and 10 years after surgery
  The Reduced WOMAC is a truncated version of the Western Ontario and McMaster's University Osteoarthritis Index. The questionnaire is designed to assess pain, disability and joint stiffness in the osteoarthritis patient.
Knee injury and Osteoarthritis Outcome Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year, 2 years, 5 years, and 10 years after surgery
  The KOOS or Knee injury and Osteoarthritis Outcome Score are patient completed questionnaires which assess the patient's opinion regarding their knee and its associated osteoarthritis.
EQ-5D | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year, 2 years, 5 years, and 10 years after surgery
  The EQ-5D is a standardized instrument for use as a measure of health outcome.
Forgotten Joint Score | 1-2 weeks prior to surgery, 1-2 weeks after surgery, 4-6 weeks after surgery, 10-12 weeks after surgery, 6 months after surgery, 1 year, 2 years, 5 years, and 10 years after surgery
  The Forgotten Joint Score is a 12-item questionnaire completed by the patient to determine how aware they are of their joint in their everyday life.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Borus, MD, Principal Investigator — Northwest Surgical Specialists / Rebound Orthopedics and Neurosurgery; Donald Roberts, MD, Principal Investigator — Northwest Surgical Specialists / Rebound Orthopedics and Neurosurgery
Locations (1):
- Rebound Orthopedics and Neurosurgery, Vancouver, Washington, United States